CLINICAL TRIAL: NCT00608530
Title: Telehealth Outreach for Chronic Back Pain
Acronym: TELE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B4767-I
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Pain; Back Pain
Keywords: pain; chronic pain; chronic back pain; randomized clinical trial
MeSH Terms: conditions — Pain; Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive Behavioral Therapy-Psychologist-Delivered (Experimental): 10 hours of Cognitive Behavioral Training delivered by a psychologist over 8 weeks by telephone and face-to-face contact
  Interventions: Behavioral: Cognitive Behavioral Therapy-Psychologist-Delivered
- Supportive Psychotherapy-Psychologist-Delivered (Active Comparator): 10 hours of Rogerian Psychotherapy delivered by a psychologist over 8 weeks by telephone and face-to-face contact
  Interventions: Behavioral: Supportive Psychotherapy-Psychologist-Delivered
- Cognitive Behavioral Therapy-Nurse-Delivered (Experimental): 10 hours of Cognitive Behavioral Training delivered by a primary care medical nurse over 8 weeks by telephone and face-to-face contact
  Interventions: Behavioral: Cognitive Behavioral Therapy Nurse-Delivered
- Supportive Psychotherapy-Nurse-Delivered (Active Comparator): 10 hours of Rogerian Psychotherapy delivered by a primary care medical nurse over 8 weeks by telephone and face-to-face contact
  Interventions: Behavioral: Supportive Psychotherapy-Nurse-Delivered

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Psychologist-Delivered — Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms; treatment was delivered by a psychologist
  Arms: Cognitive Behavioral Therapy-Psychologist-Delivered
Behavioral: Supportive Psychotherapy-Psychologist-Delivered — Supportive Psychotherapy was based on Rogerian Therapy techniques. Rogerian therapy encourages self-identification of goals and solutions using a supportive but not didactic approach; it was administered by a psychologist
  Arms: Supportive Psychotherapy-Psychologist-Delivered
Behavioral: Cognitive Behavioral Therapy Nurse-Delivered — Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms; treatment was delivered by a nurse
  Arms: Cognitive Behavioral Therapy-Nurse-Delivered
Behavioral: Supportive Psychotherapy-Nurse-Delivered — Supportive Psychotherapy was based on Rogerian Therapy techniques. Rogerian Therapy encourages self-identification of goals and solutions using a supportive but not didactic approach; it was delivered by a nurse
  Arms: Supportive Psychotherapy-Nurse-Delivered

SUMMARY:
Two separate double double blind, randomized, parallel groups, two-arm, 8 week clinical trials with 6-moth follow-up were conducted using identical inclusion/exclusion criteria and assessment batteries. In both studies patients had chronic low back pain of non-neoplastic origin. In both studies patients were randomized to one of two conditions, either a Cognitive Behavioral-based Therapy or a control condition, a supportive (Rogerian) psychotherapy. Both the cognitive-behavioral and supportive psychotherapy conditions consisted of home-based, telephone supported treatment, with 10 hours of contact time delivered over 8 weeks. In the first study (Study 1) the behavioral and Rogerian interventions were delivered by a licensed psychologist. In the second (Study 2) the interventions were delivered by a medical primary care nurse.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a major medical problem for the VA, affecting up to 15% of all veterans in primary care. Furthermore, prior surveys indicate CLBP is a leading cause of medical discharge of active duty personnel, and of medical disability costs. Given current demands on military personnel it is likely the burden of chronic pain will increase. The VA has adopted the Agency for Health Care Policy and Research Guidelines for evaluation of back pain but these guidelines do not provide specifics for true rehabilitation. It is acknowledged that most back pain patients are not surgical candidates, that medications provide only limited analgesia, and that symptom control and improved function require a comprehensive approach addressing the cognitive, affective, and behavioral aspects of chronic pain. Fortunately, structured, specific interventions to both address the multidimensional nature of pain and operationalize treatment principles in primary care settings are available. These interventions, which reflect the VA emphasis on patient-centered care, can be effective in reducing disability and pain, but are a frequently overlooked component of effective care. One reason is that most clinics lack appropriately trained psychologists. Moreover, even when specialists are available, the prevailing clinic-based service model is either too resource-intensive, or presents barriers to access.

One approach to addressing some these barriers is the use of "telehealth" outreach. Studies in diverse medical disorders and some chronic pain syndromes suggest that care can be delivered efficiently and effectively with minimal therapist contact in home-based treatment models, using telephone consultation to replace clinic visits. These approaches are fully congruent with recent VA telehealth initiatives to improve access and cost efficiency. In VA Pain Clinic settings our face-to-face, 8-week, 8-hours contact time Cognitive Behavioral Self-Management Skills Training (CBSST) program appears to be effective in reducing disability and pain, and improving mood in chronic back pain. Given the scarcity of specialized psychologists, a second approach is to train non-specialists (eg, primary care medical nurse personnel) instead of psychologists to deliver treatment, to help improve access to the intervention.

We conducted two double blind, randomized assignment, two-arm, parallel groups, six-month clinical trials. Patients with CLBP were recruited from VA San Diego primary care clinics and the community. Participants received either CBSST or Rogerian Psychotherapy in a home-based, telephone- delivered format for a total of 10 hours of therapist contact time. The methodological difference between the two studies was the discipline of the interventionist. In Study 1 the intervention was delivered by a psychologist with specific training in cognitive behavioral therapy; in Study 2 the intervention was was done by a medical primary care nurse who had been trained to deliver a version of CBSST modified to be suitable for delivery by an individual without specific expertise in cognitive behavioral therapy. The control condition was a supportive psychotherapy, again suitably modified in the case of the medical nurse interventionist. Assessments were conducted at baseline and at end of treatment, and at one, three and six months post-treatment. The primary data analytic strategy was an intent-to-treat analysis (last observation carried forward) of all participants as randomized. The primary end point was physical function (Roland & Morris Disability) at end of 8-week treatment; secondary end points were pain intensity (Numeric Rating Scale) and patient-reported clinical global impression of change. The aim of the research was to develop more accessible and more cost-efficient back pain treatment.

Key Words: Back Pain, Cognitive-Behavioral Treatment, Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75 inclusive;
2. chronic musculoskeletal low back pain (pain "on a daily basis" for at least six months) as the primary pain problem;
3. not eligible for back surgery;
4. presently lives in the San Diego area and will do so six months after baseline examination;
5. English-speaking, literate, with stable residence and phone.

Exclusion Criteria:

1. Major medical illness (e.g., insulin-dependent diabetes mellitus with neuropathy or "poor control", heart disease with New York Heart Association Functional Class III or IV, or chronic obstructive pulmonary disease requiring supplemental oxygen which might confound effects of pain on function);
2. candidate for spine surgery;
3. back pain associated with pregnancy, rheumatoid arthritis, neoplastic disease, osteomyelitis, or neural arch lesions, since their treatment and prognosis differs from the usual back pain population, or spinal stenosis, since increased physical activity would be contraindicated;
4. history of Diagnostic and Statistical Manual (DSM)-IV bipolar disorder, dementia, or schizophrenia;
5. current active DSM-IV diagnosed alcohol or non-prescribed substance dependence;
6. current active DSM-IV major depressive episode or post-traumatic stress disorder since specialty mental health care would be indicated;
7. non-opioid and opioid analgesics are permitted, except we will exclude patients on a hospital-initiated opioid treatment "contract," since at this medical center "contracting" identifies patients with history of opioid diversion, multiple VA and non-VA opioid prescribers, and repeated dose escalation in the absence of evidence of disease progression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-03; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H. Atkinson, MD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Study 1 (Psychologist-delivered treatment) recruitment commenced July 1, 2008 and concluded December 31, 2011. In Study 2 (Nurse- delivered treatment) recruitment commenced July 1, 2012 and concluded December 31, 2015. In both studies patients were recruited from VA clinics via flyers, by community newsprint advertisement, and by word of mouth.
Pre-assignment Details: In both Study 1 (Psychologist-delivered treatments, N = 66) and Study 2 (Nurse-delivered treatments, N = 67) participants who qualified and enrolled were randomized to their group assignment within 7-10 days of qualification.
Groups:
- Cognitive Behavioral Therapy-Psychologist-Dellivered: 10 hours of Cognitive Behavioral Training delivered by a psychologist over 8 weeks by telephone and face-to-face contact
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms
- Supportive Psychotherapy-Psychologist-Delivered: 10 hours of Rogerian Supportive Psychotherapy delivered by a psychologist over 8 weeks by telephone and face-to-face contact
  Rogerian supportive psychotherapy: Rogerian therapy encourages self-identification of goals and solutions using a supportive but not didactic approach
- Cognitive Behavioral Therapy-Nurse-Delivered: 10 hours of Cognitive Behavioral Training delivered by a primary care medical nurse over 8 weeks by telephone and face-to-face contact
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms
- Supportive Psychotherapy-Nurse-Delivered: 10 hours of Supportive Psychotherapy delivered by a primary care medical nurse over 8 weeks by telephone and face-to-face contact
Period: Study 1 Psychologist-delivered Treatment
Arm/Group | Cognitive Behavioral Therapy-Psychologist-Dellivered | Supportive Psychotherapy-Psychologist-Delivered | Cognitive Behavioral Therapy-Nurse-Delivered | Supportive Psychotherapy-Nurse-Delivered
Started | 33 (Randomized) | 33 (Randomized) | 0 | 0
Attended > 0 Treatment Sessions | 28 | 31 | 0 | 0
Completed | 22 | 28 | 0 | 0
Not Completed | 11 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 0 | 0
Period: Study 2 Nurse-delivered Treatments
Arm/Group | Cognitive Behavioral Therapy-Psychologist-Dellivered | Supportive Psychotherapy-Psychologist-Delivered | Cognitive Behavioral Therapy-Nurse-Delivered | Supportive Psychotherapy-Nurse-Delivered
Started | 0 | 0 | 33 | 34
Attended > 0 Treatments | 0 | 0 | 30 | 31
Completed | 0 | 0 | 21 | 27
Not Completed | 0 | 0 | 12 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3
Not completed — Lack of Efficacy | 0 | 0 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Time demands of study | 0 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ln Study 1 (Psychologist-delivered treatment) all eligible individuals who were enrolled and randomized to treatment were analyzed. In Study 2 (Nurse-delivered treatment) all participants who were randomized and attended at least 1 treatment session were analyzed.
Groups:
- Cognitive Behavioral Therapy-Psychologist-Delivered: 10 hours of Cognitive Behavioral Training delivered over 8 weeks by telephone and face-to-face contact by a psychologist
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms (e.g., pain) and set specific goals for functioning (e.g., walking 30 minutes daily).
- Supportive Psychotherapy-Psychologist-Delivered: 10 hours of Rogerian Psychotherapy delivered over 8 weeks by telephone and face-to-face contact by a psychologist
  Rogerian psychotherapy: Rogerian therapy encourages self-identification of goals and solutions using a supportive but not directive approach
- Cognitive Behavioral Therapy-Nurse-Delivered: 10 hours of Cognitive Behavioral Training delivered over 8 weeks by telephone and face-to-face contact by a medical nurse
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms (e.g., pain) and set specific goals for functioning (e.g., walking 30 minutes daily).
- Supportive Psychotherapy-Nurse-Delivered: 10 hours of Rogerian Psychotherapy delivered over 8 weeks by telephone and face-to-face contact by a medical nurse
  Rogerian psychotherapy: Rogerian therapy encourages self-identification of goals and solutions using a supportive but not directive approach
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy-Psychologist-Delivered | Supportive Psychotherapy-Psychologist-Delivered | Cognitive Behavioral Therapy-Nurse-Delivered | Supportive Psychotherapy-Nurse-Delivered | Total
Number analyzed (Participants) | 33 | 33 | 30 | 31 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.5) | 54.0 (14.8) | 62.5 (11.3) | 64.3 (12.7) | 53.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 4 | 2 | 31
  Male | 21 | 20 | 26 | 29 | 96
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 30 | 31 | 59

OUTCOME MEASURES:

1. Primary Outcome: Roland and Morris Disability Questionnaire Psychologist-Delivered Treatment Study
Description: The Roland and Morris is a 24-item self-report measure of interference of back pain on everyday function at the present time. Each item is qualified by the phrase "because of my back pain" (e.g., "Because of my back I walk more slowly than usual . . . ; Because of my back I lie down to rest more often"). Scoring the measure involves summing the number of items endorsed (from 0 to 24). Lower scores indicate less disability.
Time Frame: Baseline, End of Treatment (8 weeks)
Population: Per protocol population. All participants with baseline and Week 8 disability scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy Psychol-Delivered Treatment Study: 10 hours of Cognitive Behavioral Training delivered over 8 weeks by telephone and face-to-face contact
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms (e.g., pain) and set specific goals for functioning (e.g., walking 30 minutes daily).
- Supportive Psychotherapy-Psychologist-Delivered: 10 hours of Rogerian Psychotherapy delivered over 8 weeks by telephone and face-to-face contact
  Rogerian psychotherapy: Rogerian therapy encourages self-identification of goals and solutions using a supportive but not directive approach
Arm/Group | Cognitive Behavioral Therapy Psychol-Delivered Treatment Study | Supportive Psychotherapy-Psychologist-Delivered
Number analyzed (Participants) | 33 | 33
units on a scale
  Baseline Roland and Morris Disability | 10.0 (4.7) | 10.4 (4.4)
  Week 8 Roland and Morris Disability | 7.6 (5.0) | 7.8 (5.0)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy Psychol-Delivered Treatment Study vs Supportive Psychotherapy-Psychologist-Delivered; Repeated measures analysis of variance compared differences between and within groups (CBT and Supportive Care) from baseline to end of treatment. Statistical testing was performed using 2-tailed tests and alpha level of .05 for declaring statistical significance. The trial was powered at the >.80 level to detect differences between condition based on projected sample N = 130; given the N = 66 actually achieved our a priori power for detecting differences between groups was .63; Test type: Superiority or Other; p = .05, ANOVA

2. Primary Outcome: Roland and Morris Disability Questionnaire Nurse-Delivered Treatment Study
Description: as for outcome 1
Time Frame: Baseline, End of Treatment for Nurse-Delivered Treatment Study (8 weeks)
Population: All randomized participants who attended at least 1 treatment session were analyzed, with multiple imputation used to address missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy Nurse-Delivered Treatment Study: 10 hours of Cognitive Behavioral Training delivered over 8 weeks by telephone and face-to-face contact
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms (e.g., pain) and set specific goals for functioning (e.g., walking 30 minutes daily).
- Supportive Psychotherapy Nurse-Delivered Treatment Study: 10 hours of Rogerian Psychotherapy delivered over 8 weeks by telephone and face-to-face contact
  Rogerian psychotherapy: Rogerian therapy encourages self-identification of goals and solutions using a supportive but not directive approach
Arm/Group | Cognitive Behavioral Therapy Nurse-Delivered Treatment Study | Supportive Psychotherapy Nurse-Delivered Treatment Study
Number analyzed (Participants) | 30 | 31
units on a scale
  Baseline Roland and Morris Disability | 11.4 (5.9) | 11.1 (5.4)
  Week 8 Roland and Morris Disability | 9.4 (6.1) | 9.1 (5.2)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy Nurse-Delivered Treatment Study vs Supportive Psychotherapy Nurse-Delivered Treatment Study; Primary analyses consisted of modified intent-to-treat analysis of all randomized participants who attended at least 1 treatment session, with multiple imputation to address missing data. The study was powered at 80% to detect large effect sizes (>.50SD) and alpha of .05 with a recruitment goal N = 140; with the N = 61 actually obtained, our a priori power was .55 to detect between group differences; Test type: Superiority; p = .05, ANOVA

3. Secondary Outcome: Numeric Pain Rating Scale (Numerical Rating Scale, 0-10) Psychologist-Delivered Treatment Study
Description: The Numeric Pain Rating Scale asks the patient to rate their current intensity of pain on a scale from "0" to "1 0" where "0" indicates "no pain" and "10" indicates the "worst imaginable pain."
Time Frame: Baseline, End of Treatment (8 weeks)
Population: Intent-to-treat analysis of all randomized participants, using multiple imputation to address missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy-Psychologist Delivered: 10 hours of Cognitive Behavioral Therapy delivered over 8 weeks by a psychologist
- Supportive Care Psychologist-Delivered: 10 hours of Rogerian (Supportive) Psychotherapy delivered over 8 weeks by a psychologist
Arm/Group | Cognitive Behavioral Therapy-Psychologist Delivered | Supportive Care Psychologist-Delivered
Number analyzed (Participants) | 33 | 33
units on a scale
  Current Pain Intensity (0-10) at Baseline | 5.0 (1.8) | 5.5 (1.6)
  Current Pain Intensity at Week 8 | 4.1 (1.8) | 4.1 (1.5)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Psychologist Delivered vs Supportive Care Psychologist-Delivered; Repeated measures analysis of variance comparing groups at baseline and end of treatment; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Numeric Pain Rating Scale (Numerical Rating Scale, 0-10) Nurse-Delivered Treatment Study
Description: as for outcome 3
Time Frame: Baseline, End of Treatment of Nurse-Delivered Treatment Study (8 weeks)
Population: Modified intent-to-treat analysis of all randomized participants who attended 1 or more treatment visits; multiple imputation used to address missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy Nurse-Delivered Treatment Study: 10 hours of Cognitive Behavioral Therapy delivered over 8 weeks
- Supportive Psychotherapy Nurse-Delivered Treatment Study: 10 hours of Rogerian (Supportive) Psychotherapy delivered over 8 weeks
Arm/Group | Cognitive Behavioral Therapy Nurse-Delivered Treatment Study | Supportive Psychotherapy Nurse-Delivered Treatment Study
Number analyzed (Participants) | 30 | 31
units on a scale
  Current Pain Intensity (0-10) at Baseline | 4.9 (2.1) | 5.0 (1.9)
  Current Pain Intensity at Week 8 | 4.0 (1.9) | 3.8 (2.1)

5. Secondary Outcome: Patient-rated Global Clinical Impression of Percent Change in Overall Pain and Function
Description: Participant rating of overall improvement compared to baseline in terms of back pain impact on everyday function, self-categorized as "Better," "Worse," or "About the Same." Participants then were asked to estimate the percentage of change (i.e., 0 to 100%). Participants rating themselves as "About the Same" were coded as "0%" change. The percentage of change was calculated for each Group as a whole (Cognitive Behavioral Therapy-Psychologist Delivered compared to Supportive Care Psychologist-Delivered).
Time Frame: End of Treatment (8 weeks)
Population: Intent-to-treat analysis of all randomized participants; multiple imputation was used to address missing data.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Supportive Care-Psychologist-Delivered: 10 hours of Rogerian (Supportive) Psychotherapy delivered over 8 weeks by a psychologist
Arm/Group | Cognitive Behavioral Therapy-Psychologist Delivered | Supportive Care-Psychologist-Delivered
Number analyzed (Participants) | 33 | 33
percent change | 31 (30.4) | 18.5 (22.7)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Psychologist Delivered vs Supportive Care-Psychologist-Delivered; Test type: Superiority or Other; p = .05, Fisher Exact

6. Secondary Outcome: Percentage of Participants Rating Global Impression of Change as 'Much Improved' or 'Very Much Improved'
Description: Participant self-rating of overall change compared to baseline, considering overall function and pain intensity, using a 7-point scale ranging from 'Very Much Worse' to 'Very Much Improved.' We compared the proportion of participants in each Group rating themselves as either 'Much Improved' or 'Very Much Improved.'
Time Frame: End of Treatment (8 weeks)
Population: Modified intent-to-treat analysis of all participants who attended at least 1 treatment session
Measure: Number; unit: percentage of participants
Arm/Group | Cognitive Behavioral Therapy Nurse-Delivered Treatment Study | Supportive Psychotherapy Nurse-Delivered Treatment Study
Number analyzed (Participants) | 30 | 31
percentage of participants | 39 | 27

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Cognitive Behavioral Therapy-Psychologist-Delivered; Cognitive Behavioral Therapy-Nurse-Delivered: 10 hours of Cognitive Behavioral Training delivered over 8 weeks by telephone and face-to-face contact
  Cognitive behavioral therapy: Cognitive behavioral self-management skills training actively teaches techniques to evaluate and manage symptoms
- Supportive Psychotherapy-Psychologist-Delivered; Supportive Psychotherapy Nurse-Delivered: 10 hours of Rogerian Psychotherapy delivered over 8 weeks by telephone and face-to-face contact
  Rogerian psychotherapy: Rogerian therapists encourage individuals to identify goals and solutions using a supportive, reflective, empathic approach rather than a directive or prescriptive approach
Arm/Group | Cognitive Behavioral Therapy-Psychologist-Delivered | Supportive Psychotherapy-Psychologist-Delivered | Cognitive Behavioral Therapy-Nurse-Delivered | Supportive Psychotherapy Nurse-Delivered
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/30 | 0/31

LIMITATIONS AND CAVEATS:
The small sample size and attrition limits the strength of the evidence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes